CLINICAL TRIAL: NCT03288480
Title: A Phase 1/2a Dose-Finding Study of PT-112 in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Promontory Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-112-102
Record Dates: First submitted 2017-09-11; First posted 2017-09-20 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open-label study of PT-112 in patients with relapsed or refractory MM.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PT-112 (Other): This is a single arm study of PT-112, which is administered to patients with relapsed or refractory MM
  Interventions: Drug: PT-112

INTERVENTIONS:
Drug: PT-112 — This is a single arm study

SUMMARY:
Study PT-112-102, a multicenter, open-label dose-finding and pharmacokinetic study of PT-112 in patients with relapsed or refractory multiple myeloma.

This is designed as a two-part study. In the first part of the study, cohorts of three patients (expanded to six patients in the event of a dose-limiting toxicity) will receive escalating doses of PT-112 until the MTD is reached, based on tolerability observed during the first 28 days of treatment. In the second part of the study, an expansion cohort of 14 patients will be treated at the recommended dose to confirm the tolerability of treatment and evaluate evidence of treatment efficacy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Previously diagnosed with MM requiring treatment based on IMWG diagnostic criteria;
2. Relapsed or refractory MM after adequate exposure to and therapeutic response (following IMWG response criteria) to at least one line of treatment with one or more active agents, including alkylating drugs, corticosteroids, immunomodulatory drugs (IMiD: thalidomide, lenalidomide, pomalidomide), proteasome inhibitors (bortezomib, cartilzomib), and monoclonal antibodies (daratumumab, elotuzumab, ixazomab);
3. Evaluable MM with at least one of the following: (a) serum monoclonal component ≥ 0.5 g/dL; or (b) Bence Jones (BJ) proteinuria ≥ 200 mg/24h; or (c) measurable plasmacytoma (not previously irradiated); or (d) involved serum free light chain ≥ 10 mg/dL with an abnormal free light chain ratio;
4. ECOG Performance Status (PS) 0-2;
5. Life expectancy > 3 months;
6. At least 2 weeks (or 5 half-lives, whichever is longer) wash-out since the end of previously administered experimental therapy (6 weeks if previous nitrosourea containing regimen) or 2 weeks for standard-of-care regimens. Concurrent corticosteroids are allowed provided they are administered at an equivalent prednisone dose of ≤ 10 mg/day, as prediction or blood products only;
7. Recovery from non-hematologic toxic effects of prior therapy to grade ≤ 1 (except alopecia) by NCI CTCAE Version 4.03;
8. Adequate bone marrow (BM), renal, hepatic and metabolic function.

Key Exclusion Criteria:

1. Any of the following concomitant diseases/conditions:

   * History or presence of myocardial infarction, clinically relevant valvular heart disease, or congestive heart failure within the last 12 months;
   * Unstable cardiac dysrhythmias or persistent prolongation of the corrected QT interval (QTc) (Fridericia) to >480 msec for males or >500 msec for females, based on ECG at screening (patients with stable atrial fibrillation on treatment are allowed provided they do not meet any other cardiac or prohibited drug exclusion criterion);
   * Presence of current angina;
   * Active uncontrolled infection;
   * Morphological or cytological features of myelodysplasia and/or post-chemotherapy aplasia on BM assessment;
   * Myopathy > grade 2 or any clinical situation that causes significant and persistent elevation of CPK (>2.5 x ULN in two different determinations performed one week apart);
   * Peripheral neuropathy > grade 1, except for grade 2 without limitations on instrumental daily life activities;
   * POEMS syndrome or active plasma cell leukemia;
   * Chronic graft versus host disease (GVHD) or on immunosuppressive therapy for the control of GVHD;
   * History or presence within the last 3 months of Deep Vein Thrombosis (DVT) or a pulmonary embolism (PE);- Uncontrolled leptomeningeal disease;
   * Uncontrolled disease-related metabolic disorder (e.g., hypercalcemia);
   * Acute or chronic infections requiring systemic therapy, including, among others:
   * active infection requiring systemic therapy;
   * history of testing positive to human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome;
   * hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test is positive);
   * active tuberculosis (history of exposure or history of positive TB test with presence of clinical symptoms, physical or radiographic finding);
   * Any other major illness that, in the Investigator's judgment, may substantially increase the risk associated with the patient's participation in this study;
2. History of prior malignancy other than those previously treated with a curative intent more than 5 years ago and without relapse (any tumor) or basal cell skin cancer, in situ cervical cancer, superficial bladder cancer, or high grade intestinal polyps treated adequately, regardless of the disease-free interval;
3. Prior irradiation to > 30% of BM reserves (including total body irradiation), regardless of the washout period;
4. High dose chemotherapy followed by autologous stem cell transplantation within 90 days prior to initiating study treatment;
5. Bisphosphonate treatment within 7 days prior to initiating study treatment (while on study, bisphosphonates can be administered only once a month, between Days 18 to 21 of the 28-day treatment cycle)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Recommended dose (RD) of PT-112 for further studies in patients with relapsed or refractory multiple myeloma (MM) | 18 months

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 18 months
Area under the plasma concentration versus time curve (AUC) | 18 months
Dose-limiting toxicities (DLTs) | 18 months
Number of patients with Adverse Events (AEs) | 18 months
  Characterization of the type, incidence, severity, duration, reversibility and relationship to treatment of adverse events (AEs), and effects on vital signs and laboratory parameters.
Tumor response, including assessment of minimal residual disease, according to the International Myeloma Working Group (IMWG) response criteria | 18 months
Duration of response | 18 months
Progression free survival | 18 months
Relationship between sensitivity/response to treatment and disease status including cytogenetic biomarkers | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Leif Bergsagel, MD, Principal Investigator — Mayo Clinic
Locations (7):
- United States (7):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Oncology San Antonio Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided